CLINICAL TRIAL: NCT05690581
Title: A Nonrandomized, Open-label, Multicenter, Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Efficacy of CM369 in Subjects with Advanced Solid Tumors and Hematologic Malignancies
Brief Title: Safety, Tolerability, Pharmacokinetic Characteristics, and Efficacy of CM369 in Advanced Solid Tumors & Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM369-001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors and Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CM369 Ia Dose Escalation (Experimental): Dose escalation of CM369 as monotherapy
  Interventions: Drug: CM369
- CM369 Ib Dose Expansion (Experimental): Dose expansion of CM369 as monotherapy
  Interventions: Drug: CM369

INTERVENTIONS:
Drug: CM369 — Specified dose on specified days.

SUMMARY:
This is a nonrandomized, open-label, multicenter, phase I clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics, and efficacy of CM369 in subjects with advanced solid tumors and Hematologic Malignancies.

ELIGIBILITY:
Inclusion Criteria:

Solid tumor Inclusion Criteria:

1. Life expectancy ≥12 weeks.
2. Eastern Cooperative Oncology Group performance status of 0-1.
3. Subjects with cytology and/or histologically confirmed locally advanced unresectable or metastatic solid tumors.
4. Agree to provide archived tumor tissue samples of primary or metastatic lesions.
5. Phase Ia: have at least one measurable lesion or one evaluable lesion according to RECIST 1.1.
6. Have adequate organ function as described in the protocol.

Hematologic Malignancies Inclusion Criteria:

1. Male and female subjects ≥18 years of age and ≤ 75 years of age.
2. This study enroll subjects with recurrent/refractory hematological tumors.
3. The subjects must have measurable lesions.
4. Positive CCR8in tumor tissues of subjects.
5. Eastern Cooperative Oncology Group performance status (ECOG) of ≤2, and had a Life expectancy of at least 3 months.
6. Adequate hematological function, defined as protocol.
7. Subjects with normal coagulation function, defined as protocol.
8. Adequate hepatic, renal and cardiac functions, defined as protocol.
9. Subjects voluntarily signed informed consent form (ICF) and written informed consent must be obtained prior to performing any study-related procedure.
10. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to receiving the first dose of study medication.
11. WOCBP or male subjects and their female partners of childbearing potential must be willing to use an appropriate method of contraception during the study and for 6 months after the last dose, and must not donate eggs or sperms during this period.
12. Female subjects were not allowed to breastfeed during the study and for at least 6 months after the last dose of study medication.

Exclusion Criteria:

Solid tumor Exclusion Criteria:

1. Subjects with primary central nervous system (CNS) tumors or unstable CNS metastases.
2. Subjects who have uncontrollable or major cardiovascular disease refer to protocol.
3. Subjects who have an active autoimmune disease or have had an autoimmune disease with risk of recurrence.
4. Subjects who have active or history of interstitial lung disease or non-infectious pneumonia.
5. Subjects with any active infection requiring systemic treatment by intravenous infusion within 14 days prior to the first administration of the study drug.
6. HIV infection; Hepatitis C virus (HCV) antibody positive; HCV infection.
7. History of active bleeding within 2 months before screening, or bleeding symptoms associated with application of anticoagulant drugs or other interventions.
8. Have not recovered to CTCAE Grade 1 or better from the adverse events due to previous cancer therapies.
9. Subjects who received systemic immunosuppressive drugs within 14 days prior to the first administration of the study drug.
10. Subjects who require systemic treatment of corticosteroids or other immunosuppressive agents within 14 days prior to first dose.
11. Has a history of severe allergic reactions to monoclonal antibodies.
12. Subjects with any mental or cognitive impairment that may limit their understanding, implementation.

Hematologic Malignancies Exclusion Criteria:

1. Previous treatment with immune checkpoint inhibitors
2. Autologous hematopoietic stem cell transplantation within 100 days prior to first investigational medications dose, or history of allogeneic hematopoietic stem cell transplantation.
3. Subjects currently suffering from acute graft-versus-host disease (GVHD) or active chronic GVHD.
4. Have had any therapy directed against the subject's underlying cancer within 28 days prior to first investigational medications dose.
5. Received other clinical trial drugs within 28 days prior to first investigational medications dose.
6. Subjects who experienced major organ surgery (except for needle biopsy) or significant trauma within 28 days prior to first investigational medications administration, or who need selected surgical procedures during the study.
7. Subjects who have been vaccinated with live attenuated vaccine within 28 days prior to first investigational medications administration.
8. Clinical evidence of central nervous system (CNS) metastasis will be excluded.
9. Previous or concomitant with CNS diseases.
10. History of another primary malignancy not in remission for at least 2 years.
11. Any severe active infection requiring systemic antimicrobial therapy.
12. Active hepatitis B or C virus infection.
13. History of immunodeficiency, including human immunodeficiency virus (HIV) antibody positive or known syphilis infection.
14. History of severe cardiovascular and cerebrovascular diseases.
15. Subjects who currently or have suffered from severe interstitial lung disease.
16. The toxicity of previous anti-tumor therapy is still ≥ grade 2 at enrollment.
17. History of severe bleeding disorders,.
18. Known alcohol or drug dependence.
19. Subjects with mental disorders or poor compliance.
20. Pregnant or lactating female subjects.
21. Any other condition that, in the opinion of the investigator or project clinician, would interfere with a subject's ability to receive or complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | 90 weeks
Serious Adverse events (SAEs) | 90 weeks
Dose limiting toxicities (DLTs) | 90 weeks

SECONDARY OUTCOMES:
PK parameter: Peak Time (Tmax) | 90 weeks
PK parameter: Half-life (t1/2) | 90 weeks
PK parameter: Area Under the Curve (AUC) | 90 weeks
PK parameters: Clearance (CL) | 90 weeks
PK parameter: Apparent volume of distribution of steady state (Vss) | 90 weeks
Immunogenicity: Incidence of anti-CM369 antibody | 90 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Jilin Cancer Hospital, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No